CLINICAL TRIAL: NCT05216055
Title: Effect of Laparoscopic-Guided Transversus Abdominus Plane (TAP) Block on Opioid Consumption Using Dual-Adjunct Therapy With Dexmedetomidine and Dexamethasone Versus Liposomal Bupivacaine (Exparel®) Following Minimally Invasive Colorectal Surgery: A Single-Blinded Randomized Clinical Trial.
Brief Title: Transverse Abdominus Plane Block Study
Acronym: TAP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Accrual. PI left Institution
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-2574.cc
Record Dates: First submitted 2022-01-04; First posted 2022-01-31 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Disorders; Surgery
Keywords: Benign; Malignant; Laparoscopic Surgery; Robotic Surgery; Hybrid Surgery
MeSH Terms: interventions — Ropivacaine; Dexmedetomidine; dexamethasone 21-phosphate; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study is a randomized single blinded trial to minimize bias and provide highest level of evidence in use as part of effort to reduce opioid use consumption. This study cannot be performed as a double blinded RCT due to Exparel being milky white color in appearance and cannot be altered or shielded from being visible by the operating surgeon performing the TAP block.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Arm (Experimental): The study drug volume, concentration, and dose of treatment arm #1 selected is based on the Principal Investigator's prior experience recommendations by the Food Drug Administration (FDA), and evidence based on prior literature. The final concentration of ropivacaine is 0.375% and final volume of the mixture is 60mL.
  1. Ropivacaine 0.5% HCl, 40 mL (5 mg per mL) (200 mg)
  2. Dexmedetomidine HCl, 0.50 ml (100 ug per mL) (50 ug)
  3. Dexamethasone sodium phosphate, 1 mL (10 mg per mL) (10 mg)
  4. Normal saline 0.9%, 18.5mL
  Interventions: Combination Product: Ropivacaine, Dexmedetomidine, Dexamethasone sodium phosphate, Normal saline
- Liposomal Bupivacaine (Exparel) (Active Comparator): The study drug for patients in the treatment arm #2 will be a mixture of liposomal bupivacaine and bupivacaine 0.25% as follows:
  1. Liposomal bupivacaine, 20 mL (13.3 mg/ml) (266 mg)
  2. Normal saline 0.9%, 40mL The total volume to be injected in each patient will be 60 mL (see below for different treatment arms).
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Combination Product: Ropivacaine, Dexmedetomidine, Dexamethasone sodium phosphate, Normal saline — Ropivacaine 0.5% HCl, 40 mL (5 mg per mL) (200 mg) Dexmedetomidine HCl, 0.50 ml (100 ug per mL) (50 ug) Dexamethasone sodium phosphate, 1 mL (10 mg per mL) (10 mg) Normal saline 0.9%, 18.5mL
  Arms: Investigational Arm
Drug: Liposomal bupivacaine — Liposomal bupivacaine, 20 mL (13.3 mg/ml) (266 mg) Normal saline 0.9%, 40mL
  Other Names: Exparel
  Arms: Liposomal Bupivacaine (Exparel)

SUMMARY:
Study the effect of laparoscopic guided TAP block on opioid consumption and associated costs using a mixture of dexmedetomidine, dexamethasone, and ropivacaine versus Liposomal bupivacaine (Exparel®) in patients who undergo elective minimally invasive colorectal surgery.

DETAILED DESCRIPTION:
This is a non-inferiority single-blinded randomized trial aiming to study the effect of laparoscopic guided TAP block on opioid consumption and associated costs using a mixture of dexmedetomidine, dexamethasone, and ropivacaine versus Liposomal bupivacaine (Exparel®) in patients who undergo elective minimally invasive colorectal surgery. This study aims to continue improving our current hospital wide effort in reducing opioid consumption and, consequently, the acute and long-term consequences of opioids. It will also complement the current ongoing efforts of the Department of Surgery's quality and safety improvement project in opioid stewardship. Additionally, this dual adjunct TAP solution combination is inexpensive ($28 per injection) and may result in a significant cost savings for the hospital.

ELIGIBILITY:
Inclusion Criteria:

* provision to sign and date the consent form.
* stated willingness to comply with all study procedures and be available for the duration of the study.
* Male and female patients aged 18 and older
* Benign or malignant colorectal disease undergoing laparoscopic, robotic, or a "hybrid" (minimally invasive dissection with a 6-8 cm incision to complete the surgery) colorectal resection with or without an ostomy

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Medical conditions that may interfere with the use of the study medications (e.g., drug allergy),
* Patients with opioid dependence defined as chronic opioid use more than 3 times per week preoperatively
* Incarcerated individuals
* Age less than 18 years-old
* Urgent/emergent operations as defined by need for operation within 24 hours
* Other conditions or general disability or infirmity that in the opinion of the investigator precludes further participation in the study.
* Enrollment in another concurrent study with use of investigational drugs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Post-operative opioid consumption in the first 72 hours | 72 hours
  Total amount of both intravenous and oral opioid use in the first 72 hours after surgery measured in morphine milligram equivalents.
Post-operative opioid consumption over hospital stay | 2 months
  Total morphine dose equivalents administered throughout hospital stay
Visual analog scale pain scores in the PACU | 72 hours
  Visual analog scale (VAS) pain scores in the PACU
Visual analog scale pain scores 12 hours post op | 12 hours
  Visual analog scale pain scores 12 hours post op
Visual analog scale pain scores 24 hours post op | 24 hours
  Visual analog scale pain scores 24 hours post op
Visual analog scale pain scores 36 hours post op | 36 hours
  Visual analog scale pain scores 36 hours post op
Visual analog scale pain scores 48 hours post op | 48 hours
  Visual analog scale pain scores 48 hours post op
Visual analog scale pain scores 72 hours post op | 72 hours
  Visual analog scale pain scores 72 hours post op
Epidural need | 2 months
  Need for an epidural post-operatively. Reviewed using the EMR.
Need for postoperative patient-controlled analgesia (PCA) | 72 hours
  Determined by review of EMR. Patients use or non-use of PCA.
Need for adjunctive systemic nonopioid pain medications | 2 months
  Adjunctive systemic nonopioid pain medications
Prescribed opioid at discharge | 2 months
  Amount of opioid prescribed at discharge
Outpatient narcotic refill | 2 months
  Use the EMR to determine outpatient narcotic refill

SECONDARY OUTCOMES:
Length of hospital stay | 2 months
  To assess the impact of laparoscopic guided TAP blocks and dual-adjunct therapy on length of hospital stay following minimally invasive (laparoscopic or robotic) surgery of the colon and rectum. Calculating the length of hospital stay will allow for evaluation of effectiveness of dual adjunct therapy in context of ERAS protocol compared to liposomal bupivacaine
Use of antiemetics in the first 12 hours post op | 12 hours
  To assess the impact of laparoscopic guided TAP blocks and dual-adjunct therapy on return of bowel function following minimally invasive (laparoscopic or robotic) surgery of the colon and rectum. Antiemetic dosage reviewed using the EMR.
Use of antiemetics in the first 24 hours post op | 24 hours
  To assess the impact of laparoscopic guided TAP blocks and dual-adjunct therapy on return of bowel function following minimally invasive (laparoscopic or robotic) surgery of the colon and rectum. Antiemetic dosage reviewed using the EMR.
Use of antiemetics in the first 36 hours post op | 36 hours
  To assess the impact of laparoscopic guided TAP blocks and dual-adjunct therapy on return of bowel function following minimally invasive (laparoscopic or robotic) surgery of the colon and rectum. Antiemetic dosage reviewed using the EMR.
Use of antiemetics in the first 48 hours post op | 48 hours
  To assess the impact of laparoscopic guided TAP blocks and dual-adjunct therapy on return of bowel function following minimally invasive (laparoscopic or robotic) surgery of the colon and rectum. Antiemetic dosage reviewed using the EMR.
Use of antiemetics in the first 72 hours post op | 72 hours
  To assess the impact of laparoscopic guided TAP blocks and dual-adjunct therapy on return of bowel function following minimally invasive (laparoscopic or robotic) surgery of the colon and rectum. Antiemetic dosage reviewed using the EMR.
Time to first flatus | 2 months
  Days from surgery to first flatus postoperatively. Reviewed using the EMR.
Time to first bowel movement | 2 months
  Days from surgery to first bowel movement postoperatively. Reviewed using the EMR.
Need to insert nasogastric tube | 2 months
  To assess the impact of laparoscopic guided TAP blocks and dual-adjunct therapy on return of bowel function following minimally invasive (laparoscopic or robotic) surgery of the colon and rectum. Reviewed using the EMR.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon C Chapman, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No